CLINICAL TRIAL: NCT05464134
Title: Incidence of Lumbar Spondylolisthesis in Patients Candidate for Total Knee Replacement
Brief Title: Incidence of Lumbar Spondylolisthesis in Patients Candidate for TKR
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Mario Sameh Wadie Narouz, Principal Investigator, Assiut University
Other Study IDs: Lumbar Spondylolisthesis & TKR
Record Dates: First submitted 2022-05-27; First posted 2022-07-19 (Actual); Last update posted 2023-05-19 (Actual); Status verified 2023-05

CONDITIONS: Lumbar Spondylolisthesis
MeSH Terms: conditions — Spondylolisthesis | interventions — X-Rays

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Radiation: x-ray — plain radiographs of lower limb anteroposterior and lateral views , lumbar spine plain radiographs (anteroposterior, lateral, lateral in flexion and lateral in extension views )

SUMMARY:
This study aims to detect the incidence of spondylolisthesis in patients candidate for Total knee replacement (TKR) and to investigate the effect of TKR on the course of low back pain.

DETAILED DESCRIPTION:
Total Knee Replacement (TKR) is one of the most successful surgeries in modern-day orthopedics, performed mainly to treat end-stage knee osteoarthritis (OA) . degenerative spondylolisthesis is one of the most common causes of low back pain where a spinal vertebra slides from its anatomical position, affecting about 11.5% of the population, furthermore, many elderly patients undergoing TKR usually suffer from spondylolisthesis.

Spondylolisthesis with subsequent lumbar spine degenerative disease presents as lower back and radiating pain to the legs at rest or during activity, Spondylolisthesis causes hamstring tightness which is felt as pain at the back of the knee, lumbar radiculopathy of the L3 root nerve could vary from thigh pain to hip and/or knee pain, all of which could be misled as pain due to knee OA . On the other hand, patients having knee OA with a flexion deformity compensate their posture by increasing the lumbar lordosis, if the lumbar spine lost its ability to compensate for the knee deformity, this could aggravate low back pain and enhance further lumbar spine instability and spondylosis .

In addition, the persistence of coexisting lumbar spine symptoms after TKA might adversely affect postoperative outcomes in terms of pain and function, even after successful TKA .

Chang et al., studied the prevalence and severity of coexisting lumbar spondylosis in terms of radiographic lumbar spine degeneration and lumbar spine symptoms in patients with advanced knee OA undergoing TKR, in their study, 51% of patients undergoing TKR had at least one moderate to severe lumbar spine symptom, and patients with severe radicular pain on the activity before the TKR was likely to demonstrate poor knee function 2 years post-TKR . This is why lumbar spine pathologies should be fully investigated in patients coming for TKR.

ELIGIBILITY:
Inclusion Criteria:

* primary end-stage knee osteoarthritis.

Exclusion Criteria:

* secondary inflammatory knee osteoarthritis.
* post traumatic knee osteoarthritis.
* patients with active infection.
* patients with poor general condition.
* patients who had previous spinal fixation or fusion surgery.

Min Age: 40 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: The sample size was calculated using STAT CALC based on the previous work by Chang et al., 2014 (4), by considering the following assumptions:- 95% two-sided confidence level, with a power of 80% & Alpha error of 5% odds ratio calculated= 1.115. The final maximum sample size was 200
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2023-05 (Estimated); Primary Completion 2024-05 (Estimated); Study Completion 2024-06 (Estimated)

PRIMARY OUTCOMES:
Incidence of lumbar spine spondylolisthesis. | Baseline
  showing the incidence and occurrence of Lumbar Spondylolisthesis in patients with severe knee Osteoarthritis which needs Total knee replacement
Severity of lumbar spine spondylolisthesis. | Baseline
  showing the grades of lumbar spine spondylolisthesis through The Meyerding classification system with grade 1 is the minimum and grade 5 is the maximum which in turn has the worst outcome
occurence of lumbar spine spondylolishtesis Occurrence of lumbar spine spondylolisthesis | Baseline
  Showing the occurrence of lumbar spine spondylolisthesis in patients with severe osteoarthritis which needs total knee replacement

SECONDARY OUTCOMES:
Change in characters of low back pain over the postoperative period. | 6 months follow up
  Recording the changes of the backpain after Total knee replacement using Oswestry disability index scale which is 0 is the minimum value and 100 is the maximum value which in turn presents with the worst outcome
Spine radiological features. | Baseline
  Recording the radiological features of Lumber spine through plain xrays of to evaluate the presence of Spondylolisthesis
Knee radiological and alignment features. | Baseline
  Recording the radiological features of knee through plain xrays of to measure the hip knee ankle angle

REFERENCES:
- [Background] Kahlenberg CA, Nwachukwu BU, McLawhorn AS, Cross MB, Cornell CN, Padgett DE. Patient Satisfaction After Total Knee Replacement: A Systematic Review. HSS J. 2018 Jul;14(2):192-201. doi: 10.1007/s11420-018-9614-8. Epub 2018 Jun 5. PMID 29983663
- [Background] Patel EA, Perloff MD. Radicular Pain Syndromes: Cervical, Lumbar, and Spinal Stenosis. Semin Neurol. 2018 Dec;38(6):634-639. doi: 10.1055/s-0038-1673680. Epub 2018 Dec 6. PMID 30522138
- [Background] Londhe SB, Shah RV, Patwardhan M, Doshi AP, Londhe SS, Subhedar K, Kundnani V, Patel J. Study of Patients with Bilateral Knee Osteoarthritis Undergoing Total Knee Replacement Procedure with Coexisting Lumbar Spondylosis Symptoms. Asian Spine J. 2021 Dec;15(6):825-830. doi: 10.31616/asj.2020.0279. Epub 2020 Dec 28. PMID 33355851
- [Background] Chang CB, Park KW, Kang YG, Kim TK. Coexisting lumbar spondylosis in patients undergoing TKA: how common and how serious? Clin Orthop Relat Res. 2014 Feb;472(2):710-7. doi: 10.1007/s11999-013-3298-7. Epub 2013 Sep 25. PMID 24065173
- See also: Decompression with or without fusion in degenerative lumbar spondylolisthesis — http://www.nejm.org/doi/full/10.1056/NEJMoa2100990